CLINICAL TRIAL: NCT05403593
Title: Registry of Emergent Large VeSsel OCclUsion DuE to IntraCranial AtherosclerosiS
Acronym: RESCUE-ICAS
Status: Completed | Type: Observational
Sponsor: Medical University of South Carolina (Other)
Collaborators: University of Göttingen (Other); Thomas Jefferson University (Other); University of Miami (Other); University of Basel (Other); University of Tennessee (Other); Wake Forest University Health Sciences (Other); Emory University (Other); The University of Texas Health Science Center at San Antonio (Other); University of Iowa (Other); Indiana University (Other); University of Chicago (Other); Careggi Hospital (Other); Massachusetts General Hospital (Other); Imam Abdulrahman Bin Faisal University (Other); Brown University (Other); Yale University (Other); Sutter Health (Other); Centro Hospitalar de Lisboa Central (Other); HCA Houston Healthcare Kingwood (Unknown); advocate christ medical center (Unknown)
Responsible Party: Principal Investigator, Sami Al Kasab, MD, Medical University of South Carolina
Other Study IDs: Pro00115854
Record Dates: First submitted 2022-05-24; First posted 2022-06-03 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-03

CONDITIONS: Intracranial Stenosis; Large Vessel Occlusion; Mechanical Thrombectomy
Keywords: Intracranial Stenosis; Large Vessel Occlusion

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants with Intracranial Stenosis: Patients with Intracranial Stenosis who undergo Mechanical Thrombectomy will be added to the registry given they meet the age inclusion criteria.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No intervention, prospective data collection

SUMMARY:
The aim of this study is to develop an international multicenter registry of patient data and outcomes for patients undergoing mechanical thrombectomy for emergent large vessel occlusion with residual underlying stenosis following successful revascularization.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing mechanical thrombectomy
* AND have intracranial stenosis
* Patients aged 18-90 years

Exclusion Criteria:

* None

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects aged 18-90 years will be identified once they undergo mechanical thrombectomy and identified as having intracranial stenosis as the etiology for large vessel occlusion.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2024-03-05 (Actual); Study Completion 2024-06-14 (Actual)

PRIMARY OUTCOMES:
modified Rankin score | pre-stroke
  standard stroke score measuring disability level delivered by physician with level 0-6 with 0 being no symptoms and 6 being death. Outcome measured by the distribution of mRS score.
modified Rankin score | 7 days
  standard stroke score measuring disability level delivered by physician with level 0-6 with 0 being no symptoms and 6 being death. Outcome measured by the distribution of mRS score.
modified Rankin score | admission
  standard stroke score measuring disability level delivered by physician with level 0-6 with 0 being no symptoms and 6 being death. Outcome measured by the distribution of mRS score.
modified Rankin score | 3 months
  standard stroke score measuring disability level delivered by physician with level 0-6 with 0 being no symptoms and 6 being death. Outcome measured by the distribution of mRS score.
Mortality | 90 day
  Death at 90 days post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Sami Al Kasab, MD, Principal Investigator — Medical University of South Carolina
Locations (19):
- United States (14):
  - Yale New Haven Hospital, New Haven, Connecticut
  - Univeristy of Miami Health System, Miami, Florida
  - Emory Univeristy Hospital, Atlanta, Georgia
  - Univeristy of Chicago Medicine, Chicago, Illinois
  - Advocate Aurora Health, Oak Lawn, Illinois
  - Indiana Health Univeristy Hospital, Indianapolis, Indiana
  - Univeristy of Iowa Hospital, Iowa City, Iowa
  - Massachuestts General Hospital, Boston, Massachusetts
  - Atrium Health Wake Forest Baptist, Winston-Salem, North Carolina
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Brown University, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - The University of Tennessee Health Science Center, Memphis, Tennessee
  - Univeristy of Texas Health Science Center at San Antonio, San Antonio, Texas
- Universitätsmedizin Göttingen, Göttingen, Germany, Germany
- Careggi Universtiy Hospital, Florence, Florence, Italy
- Nova University Lisbon, Lisbon, Portugal, Portugal
- Imam Abdulrahman Alfaisal University, Dammam, Dammam, Saudi Arabia
- Universitätsspital Basel, Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No
All data will be de-identified

REFERENCES:
- [Background] Powers WJ, Rabinstein AA, Ackerson T, Adeoye OM, Bambakidis NC, Becker K, Biller J, Brown M, Demaerschalk BM, Hoh B, Jauch EC, Kidwell CS, Leslie-Mazwi TM, Ovbiagele B, Scott PA, Sheth KN, Southerland AM, Summers DV, Tirschwell DL. Guidelines for the Early Management of Patients With Acute Ischemic Stroke: 2019 Update to the 2018 Guidelines for the Early Management of Acute Ischemic Stroke: A Guideline for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2019 Dec;50(12):e344-e418. doi: 10.1161/STR.0000000000000211. Epub 2019 Oct 30. PMID 31662037
- [Background] Khatri P, Abruzzo T, Yeatts SD, Nichols C, Broderick JP, Tomsick TA; IMS I and II Investigators. Good clinical outcome after ischemic stroke with successful revascularization is time-dependent. Neurology. 2009 Sep 29;73(13):1066-72. doi: 10.1212/WNL.0b013e3181b9c847. PMID 19786699
- [Background] Kleine JF, Wunderlich S, Zimmer C, Kaesmacher J. Time to redefine success? TICI 3 versus TICI 2b recanalization in middle cerebral artery occlusion treated with thrombectomy. J Neurointerv Surg. 2017 Feb;9(2):117-121. doi: 10.1136/neurintsurg-2015-012218. Epub 2016 Feb 17. PMID 26888952
- [Background] Zaidat OO, Castonguay AC, Nogueira RG, Haussen DC, English JD, Satti SR, Chen J, Farid H, Borders C, Veznedaroglu E, Binning MJ, Puri A, Vora NA, Budzik RF, Dabus G, Linfante I, Janardhan V, Alshekhlee A, Abraham MG, Edgell R, Taqi MA, Khoury RE, Mokin M, Majjhoo AQ, Kabbani MR, Froehler MT, Finch I, Ansari SA, Novakovic R, Nguyen TN. TREVO stent-retriever mechanical thrombectomy for acute ischemic stroke secondary to large vessel occlusion registry. J Neurointerv Surg. 2018 Jun;10(6):516-524. doi: 10.1136/neurintsurg-2017-013328. Epub 2017 Sep 29. PMID 28963367
- [Background] Goyal M, Menon BK, van Zwam WH, Dippel DW, Mitchell PJ, Demchuk AM, Davalos A, Majoie CB, van der Lugt A, de Miquel MA, Donnan GA, Roos YB, Bonafe A, Jahan R, Diener HC, van den Berg LA, Levy EI, Berkhemer OA, Pereira VM, Rempel J, Millan M, Davis SM, Roy D, Thornton J, Roman LS, Ribo M, Beumer D, Stouch B, Brown S, Campbell BC, van Oostenbrugge RJ, Saver JL, Hill MD, Jovin TG; HERMES collaborators. Endovascular thrombectomy after large-vessel ischaemic stroke: a meta-analysis of individual patient data from five randomised trials. Lancet. 2016 Apr 23;387(10029):1723-31. doi: 10.1016/S0140-6736(16)00163-X. Epub 2016 Feb 18. PMID 26898852
- [Background] Zaidat OO, Mueller-Kronast NH, Hassan AE, Haussen DC, Jadhav AP, Froehler MT, Jahan R, Ali Aziz-Sultan M, Klucznik RP, Saver JL, Hellinger FR Jr, Yavagal DR, Yao TL, Gupta R, Martin CO, Bozorgchami H, Kaushal R, Nogueira RG, Gandhi RH, Peterson EC, Dashti S, Given CA 2nd, Mehta BP, Deshmukh V, Starkman S, Linfante I, McPherson SH, Kvamme P, Grobelny TJ, Hussain MS, Thacker I, Vora N, Chen PR, Monteith SJ, Ecker RD, Schirmer CM, Sauvageau E, Chebl AB, Derdeyn CP, Maidan L, Badruddin A, Siddiqui AH, Dumont TM, Alhajeri A, Taqi MA, Asi K, Carpenter J, Boulos A, Jindal G, Puri AS, Chitale R, Deshaies EM, Robinson D, Kallmes DF, Baxter BW, Jumaa M, Sunenshine P, Majjhoo A, English JD, Suzuki S, Fessler RD, Delgado-Almandoz J, Martin JC, Liebeskind DS; STRATIS Investigators. Impact of Balloon Guide Catheter Use on Clinical and Angiographic Outcomes in the STRATIS Stroke Thrombectomy Registry. Stroke. 2019 Mar;50(3):697-704. doi: 10.1161/STROKEAHA.118.021126. PMID 30776994
- [Background] Kaesmacher J, Gralla J, Mosimann PJ, Zibold F, Heldner MR, Piechowiak E, Dobrocky T, Arnold M, Fischer U, Mordasini P. Reasons for Reperfusion Failures in Stent-Retriever-Based Thrombectomy: Registry Analysis and Proposal of a Classification System. AJNR Am J Neuroradiol. 2018 Oct;39(10):1848-1853. doi: 10.3174/ajnr.A5759. Epub 2018 Aug 30. PMID 30166434
- [Background] Kang DH, Kim YW, Hwang YH, Park SP, Kim YS, Baik SK. Instant reocclusion following mechanical thrombectomy of in situ thromboocclusion and the role of low-dose intra-arterial tirofiban. Cerebrovasc Dis. 2014;37(5):350-5. doi: 10.1159/000362435. Epub 2014 Jun 13. PMID 24941966
- [Background] Chimowitz MI, Lynn MJ, Derdeyn CP, Turan TN, Fiorella D, Lane BF, Janis LS, Lutsep HL, Barnwell SL, Waters MF, Hoh BL, Hourihane JM, Levy EI, Alexandrov AV, Harrigan MR, Chiu D, Klucznik RP, Clark JM, McDougall CG, Johnson MD, Pride GL Jr, Torbey MT, Zaidat OO, Rumboldt Z, Cloft HJ; SAMMPRIS Trial Investigators. Stenting versus aggressive medical therapy for intracranial arterial stenosis. N Engl J Med. 2011 Sep 15;365(11):993-1003. doi: 10.1056/NEJMoa1105335. Epub 2011 Sep 7. PMID 21899409
- [Background] Zaidat OO, Fitzsimmons BF, Woodward BK, Wang Z, Killer-Oberpfalzer M, Wakhloo A, Gupta R, Kirshner H, Megerian JT, Lesko J, Pitzer P, Ramos J, Castonguay AC, Barnwell S, Smith WS, Gress DR; VISSIT Trial Investigators. Effect of a balloon-expandable intracranial stent vs medical therapy on risk of stroke in patients with symptomatic intracranial stenosis: the VISSIT randomized clinical trial. JAMA. 2015 Mar 24-31;313(12):1240-8. doi: 10.1001/jama.2015.1693. PMID 25803346
- [Background] Chimowitz MI, Lynn MJ, Howlett-Smith H, Stern BJ, Hertzberg VS, Frankel MR, Levine SR, Chaturvedi S, Kasner SE, Benesch CG, Sila CA, Jovin TG, Romano JG; Warfarin-Aspirin Symptomatic Intracranial Disease Trial Investigators. Comparison of warfarin and aspirin for symptomatic intracranial arterial stenosis. N Engl J Med. 2005 Mar 31;352(13):1305-16. doi: 10.1056/NEJMoa043033. PMID 15800226
- [Background] Yu SC, Cheng HK, Cheng PW, Lui WM, Leung KM, Tan CB, Pang KY, Wong GK, Cheung YL, Lee R, Wong YC, Wong CK, Kwok JC; Hong Kong Society of Interventional and Therapeutic Neuroradiology. Angioplasty and stenting for intracranial atherosclerotic stenosis: position statement of the Hong Kong Society of Interventional and Therapeutic Neuroradiology. Hong Kong Med J. 2013 Feb;19(1):69-73. PMID 23378358
- [Derived] Al Kasab S, Almallouhi E, Jumaa M, Inoa V, Capasso F, Nahhas M, Starke RM, Fragata I, Bender M, Moldovan K, Yaghi S, Maier I, Grossberg JA, Jabbour P, Psychogios M, Samaniego EA, Burkhardt JK, Jankowitz B, Abdalkader M, Hassan AE, Altschul D, Mascitelli J, Regenhardt RW, Wolfe S, Ezzeldin M, Limaye K, Grandhi R, Al Jehani H, Niazi M, Goyal N, Tjoumakaris S, Alawieh A, Abdelsalam A, Guada L, Ntoulias N, El-Ghawanmeh R, Batra V, Choi A, Zohdy YM, Nguyen S, Essibayi MA, El Naamani K, Koo A, Almekhlafi M, Raz E, Miller S, Mierzwa A, Zaidi S, Gudino AS, Alsarah A, Azeem HM, Mattingly TK, Schartz DA, Nelson A, Pinheiro C, Spiotta AM, Kicielinski K, Lena J, Lajthia O, Hubbard Z, Zaidat OO, Derdeyn CP, Klein P, Nguyen TN, de Havenon A. Outcomes of Adjunct Emergent Stenting Versus Mechanical Thrombectomy Alone: The RESCUE-ICAS Registry. Stroke. 2025 Feb;56(2):390-400. doi: 10.1161/STROKEAHA.124.049038. Epub 2024 Nov 22. PMID 39576761